CLINICAL TRIAL: NCT02945410
Title: Can Increased Dietary Protein Prevent the Suppression of Metabolism and Maintain Anabolic Sensitivity of Bone and Skeletal Muscle During Caloric Restriction?
Brief Title: Effect of Caloric Restriction and Protein Intake on Metabolism and Anabolic Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 15895
Record Dates: First submitted 2016-10-10; First posted 2016-10-26 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Weight Loss; Starvation
MeSH Terms: conditions — Weight Loss; Starvation | interventions — Caloric Restriction; Proteins; Exercise; Calcium; Vitamin D; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Caloric Restriction and High Protein (Experimental): Participants will be calorie restricted to 30 kcal/kg FFM/day and consume 1.7 g protein/kg BW/day.
  Interventions: Other: Caloric Restriction; Other: Protein; Other: Exercise; Dietary Supplement: Calcium and Vitamin D; Other: Maltodextrin
- Caloric Restriction and Normal Protein (Active Comparator): Participants will be calorie restricted to 30 kcal/kg FFM/day and consume 0.8 g protein/kg BW/day.
  Interventions: Other: Caloric Restriction; Other: Exercise; Dietary Supplement: Calcium and Vitamin D; Other: Maltodextrin
- Energy Balance (Placebo Comparator): Participants will be in energy balance and consume 1.7 g protein/kg BW/day.
  Interventions: Other: Protein; Other: Exercise; Dietary Supplement: Calcium and Vitamin D; Other: Maltodextrin

INTERVENTIONS:
Other: Caloric Restriction — Participants will consume 30 kcal/kg FFM/day.
  Arms: Caloric Restriction and High Protein; Caloric Restriction and Normal Protein
Other: Protein — Participants will consume 1.7 g protein/kg BW/day.
  Arms: Caloric Restriction and High Protein; Energy Balance
Other: Exercise — Participants will conduct aerobic exercise designed to expend 15 kcal/kg FFM/day
Dietary Supplement: Calcium and Vitamin D — Participants will be provided calcium and vitamin D supplement in order to maintain calcium and Vitamin D intake constant across all study arms
Other: Maltodextrin — Participants will be provided with maltodextrin to supplement the liquid diet in order to meet caloric needs within each study arm

SUMMARY:
The purpose of this study is to determine if an increased protein intake can attenuate the suppression of metabolic and anabolic hormones during caloric restriction

DETAILED DESCRIPTION:
1. Preliminary testing

   Prior to the study start, participants will be weighed and body composition will be determined using calipermetry (7 sites) and bioelectrical impedance. Peak oxygen uptake (VO2peak) will be assessed using an incremental exercise test on a bicycle ergometer.
2. Randomization

   Participants will proceed through each of the following conditions lasting 5 days:

   CR-LP: Participants will be restricted to 30 kcal/kg FFM/day and protein intake will be low (0.8 g/kg BW/day).

   CR-HP: Participants will be restricted to 30 kcal/kg FFM/day and protein intake will be high (1.7 g/kg BW/day).

   CON: Participants will be in energy balance and consume 1.7 g protein/kg BW/day.
3. Diet Prescription

   Dietary energy intake will be controlled using clinical products and maltodextrin to meet target energy intakes. Participants will received calcium and Vitamin D supplementation throughout the study.
4. Exercise Prescription

   During all conditions, participants will conduct daily supervised exercise on a bicycle ergometer at an exercise intensity of 60% VO2peak. Exercise duration will be adjusted individually such that exercise energy expenditure will amount to 15 kcal/kg FFM/day. Additional exercise and intense physical activity will be prohibited.
5. Assessments

   The following assessments will be conducted prior to the start of each condition as well as upon completion of each condition: body weight and composition (impedance), fasting blood draw for assessment of metabolic and anabolic hormones, resting metabolic rate, aerobic fitness (VO2peak), and questionnaires.
6. Washout

Once a participant has completed a study condition, participant will be allowed a washout of at least 14 days to allow protein balance to return to baseline (Hoffer & Forse, 1990). During this time, participants will resume their regular diet and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 4 hours/week of purposeful aerobic exercise over the last 3 months
* Body mass index: 19-25 kg/m2
* < 15% body fat

Exclusion Criteria:

* Cardiovascular disease risk factors that would result in greater than low risk
* Smoking
* Type I, type II diabetes, or history of high fasting glucose;
* History of high blood pressure and/or use of medication for hypertension;
* History of Dyslipidemia, or on lipid-lowering medication;
* Underlying health condition and/or use of medication that could interfere with any of our study outcomes.
* History or current diagnosis of a clinical eating disorder
* Failure to adhere to study protocol

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Koehler, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- Sports and Exercise Nutrition Laboratory, Department of Nutrition and Health Sciences, Ruth Leverton Hall, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill JO. Understanding and addressing the epidemic of obesity: an energy balance perspective. Endocr Rev. 2006 Dec;27(7):750-61. doi: 10.1210/er.2006-0032. Epub 2006 Nov 22. PMID 17122359
- [Background] Donnelly JE, Blair SN, Jakicic JM, Manore MM, Rankin JW, Smith BK; American College of Sports Medicine. American College of Sports Medicine Position Stand. Appropriate physical activity intervention strategies for weight loss and prevention of weight regain for adults. Med Sci Sports Exerc. 2009 Feb;41(2):459-71. doi: 10.1249/MSS.0b013e3181949333. PMID 19127177
- [Background] Weinheimer EM, Sands LP, Campbell WW. A systematic review of the separate and combined effects of energy restriction and exercise on fat-free mass in middle-aged and older adults: implications for sarcopenic obesity. Nutr Rev. 2010 Jul;68(7):375-88. doi: 10.1111/j.1753-4887.2010.00298.x. PMID 20591106
- [Background] Forbes GB. Body fat content influences the body composition response to nutrition and exercise. Ann N Y Acad Sci. 2000 May;904:359-65. doi: 10.1111/j.1749-6632.2000.tb06482.x. PMID 10865771
- [Background] Areta JL, Burke LM, Camera DM, West DW, Crawshay S, Moore DR, Stellingwerff T, Phillips SM, Hawley JA, Coffey VG. Reduced resting skeletal muscle protein synthesis is rescued by resistance exercise and protein ingestion following short-term energy deficit. Am J Physiol Endocrinol Metab. 2014 Apr 15;306(8):E989-97. doi: 10.1152/ajpendo.00590.2013. Epub 2014 Mar 4. PMID 24595305
- [Background] Carbone JW, Pasiakos SM, Vislocky LM, Anderson JM, Rodriguez NR. Effects of short-term energy deficit on muscle protein breakdown and intramuscular proteolysis in normal-weight young adults. Appl Physiol Nutr Metab. 2014 Aug;39(8):960-8. doi: 10.1139/apnm-2013-0433. Epub 2014 Jun 19. PMID 24945715
- [Background] Wasserman DH, Kang L, Ayala JE, Fueger PT, Lee-Young RS. The physiological regulation of glucose flux into muscle in vivo. J Exp Biol. 2011 Jan 15;214(Pt 2):254-62. doi: 10.1242/jeb.048041. PMID 21177945
- [Background] Gault ML, Willems ME. Aging, functional capacity and eccentric exercise training. Aging Dis. 2013 Sep 25;4(6):351-63. doi: 10.14336/AD.2013.0400351. PMID 24307968
- [Background] Dulloo AG, Jacquet J, Montani JP, Schutz Y. How dieting makes the lean fatter: from a perspective of body composition autoregulation through adipostats and proteinstats awaiting discovery. Obes Rev. 2015 Feb;16 Suppl 1:25-35. doi: 10.1111/obr.12253. PMID 25614201
- [Background] Wade GN, Schneider JE, Li HY. Control of fertility by metabolic cues. Am J Physiol. 1996 Jan;270(1 Pt 1):E1-19. doi: 10.1152/ajpendo.1996.270.1.E1. PMID 8772468
- [Background] Loucks AB. Energy balance and body composition in sports and exercise. J Sports Sci. 2004 Jan;22(1):1-14. doi: 10.1080/0264041031000140518. PMID 14974441
- [Background] Misra M, Klibanski A. The neuroendocrine basis of anorexia nervosa and its impact on bone metabolism. Neuroendocrinology. 2011;93(2):65-73. doi: 10.1159/000323771. Epub 2011 Jan 13. PMID 21228564
- [Background] Ihle R, Loucks AB. Dose-response relationships between energy availability and bone turnover in young exercising women. J Bone Miner Res. 2004 Aug;19(8):1231-40. doi: 10.1359/JBMR.040410. Epub 2004 Apr 19. PMID 15231009
- [Background] De Souza MJ, Williams NI. Beyond hypoestrogenism in amenorrheic athletes: energy deficiency as a contributing factor for bone loss. Curr Sports Med Rep. 2005 Feb;4(1):38-44. doi: 10.1007/s11932-005-0029-1. PMID 15659278
- [Background] Rizzoli R, Bianchi ML, Garabedian M, McKay HA, Moreno LA. Maximizing bone mineral mass gain during growth for the prevention of fractures in the adolescents and the elderly. Bone. 2010 Feb;46(2):294-305. doi: 10.1016/j.bone.2009.10.005. Epub 2009 Oct 17. PMID 19840876
- [Background] Pikosky MA, Smith TJ, Grediagin A, Castaneda-Sceppa C, Byerley L, Glickman EL, Young AJ. Increased protein maintains nitrogen balance during exercise-induced energy deficit. Med Sci Sports Exerc. 2008 Mar;40(3):505-12. doi: 10.1249/MSS.0b013e31815f6643. PMID 18379214
- [Background] Pasiakos SM, Margolis LM, McClung JP, Cao JJ, Whigham LD, Combs GF, Young AJ. Whole-body protein turnover response to short-term high-protein diets during weight loss: a randomized controlled trial. Int J Obes (Lond). 2014 Jul;38(7):1015-8. doi: 10.1038/ijo.2013.197. Epub 2013 Oct 29. PMID 24166063
- [Background] Chevalley T, Bonjour JP, Ferrari S, Rizzoli R. High-protein intake enhances the positive impact of physical activity on BMC in prepubertal boys. J Bone Miner Res. 2008 Jan;23(1):131-42. doi: 10.1359/jbmr.070907. PMID 17892378
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants Excluded prior to assignment:
  n = 4 did not meet inclusion criteria on preliminary questionnaires (n = 1 did not met the age requirements (reported a false age) n = 1 reported hyperthyroidism n = 2 reported insufficient levels of physical activity) n = 1 declined to participate in the study after enrolling
Groups:
- (1) CRHP (2) EB (3) CRNP: In the Caloric Restriction and High Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 1.7 g protein/kg BW/day.
  In the Energy Balance Intervention, participants will consume 55 kcal/kg FFM/day and 1.7 g protein/kg BW/day.
  In the Caloric Restriction and Normal Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 0.8 g protein/kg BW/day.
  In all Interventions, participants will conduct aerobic exercise designed to expend 15 kcal/kg FFM/day. Participants will be provided calcium and vitamin D supplement in order to maintain calcium and Vitamin D intake constant across all study arms. Participants will be provided with maltodextrin to supplement the liquid diet in order to meet caloric needs within each study arm.
- (1) CRHP (2) CRNP (3) EB: In the Caloric Restriction and High Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 1.7 g protein/kg BW/day.
  In the Caloric Restriction and Normal Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 0.8 g protein/kg BW/day.
  In the Energy Balance Intervention, participants will consume 55 kcal/kg FFM/day and 1.7 g protein/kg BW/day.
  In all Interventions, participants will conduct aerobic exercise designed to expend 15 kcal/kg FFM/day. Participants will be provided calcium and vitamin D supplement in order to maintain calcium and Vitamin D intake constant across all study arms. Participants will be provided with maltodextrin to supplement the liquid diet in order to meet caloric needs within each study arm.
- (1) CRNP (2) EB (3) CRHP: In the Caloric Restriction and Normal Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 0.8 g protein/kg BW/day.
  In the Energy Balance Intervention, participants will consume 55 kcal/kg FFM/day and 1.7 g protein/kg BW/day.
  In the Caloric Restriction and High Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 1.7 g protein/kg BW/day.
  In all Interventions, participants will conduct aerobic exercise designed to expend 15 kcal/kg FFM/day. Participants will be provided calcium and vitamin D supplement in order to maintain calcium and Vitamin D intake constant across all study arms. Participants will be provided with maltodextrin to supplement the liquid diet in order to meet caloric needs within each study arm.
- (1) CRNP (2) CRHP (3) EB: In the Caloric Restriction and Normal Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 0.8 g protein/kg BW/day.
  In the Caloric Restriction and High Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 1.7 g protein/kg BW/day.
  In the Energy Balance Intervention, participants will consume 55 kcal/kg FFM/day and 1.7 g protein/kg BW/day.
  In all Interventions, participants will conduct aerobic exercise designed to expend 15 kcal/kg FFM/day. Participants will be provided calcium and vitamin D supplement in order to maintain calcium and Vitamin D intake constant across all study arms. Participants will be provided with maltodextrin to supplement the liquid diet in order to meet caloric needs within each study arm.
- (1) EB (2) CRHP (3) CRNP: In the Energy Balance Intervention, participants will consume 55 kcal/kg FFM/day and 1.7 g protein/kg BW/day.
  In the Caloric Restriction and High Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 1.7 g protein/kg BW/day.
  In the Caloric Restriction and Normal Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 0.8 g protein/kg BW/day.
  In all Interventions, participants will conduct aerobic exercise designed to expend 15 kcal/kg FFM/day. Participants will be provided calcium and vitamin D supplement in order to maintain calcium and Vitamin D intake constant across all study arms. Participants will be provided with maltodextrin to supplement the liquid diet in order to meet caloric needs within each study arm.
- (1) EB (2) CRNP (3) CRHP: In the Energy Balance Intervention, participants will consume 55 kcal/kg FFM/day and 1.7 g protein/kg BW/day.
  In the Caloric Restriction and Normal Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 0.8 g protein/kg BW/day.
  In the Caloric Restriction and High Protein Intervention, participants will be calorie restricted to 30 kcal/kg FFM/day and consume 1.7 g protein/kg BW/day.
  In all Interventions, participants will conduct aerobic exercise designed to expend 15 kcal/kg FFM/day. Participants will be provided calcium and vitamin D supplement in order to maintain calcium and Vitamin D intake constant across all study arms. Participants will be provided with maltodextrin to supplement the liquid diet in order to meet caloric needs within each study arm.
Period: Intervention 1 (5 Days)
Arm/Group | (1) CRHP (2) EB (3) CRNP | (1) CRHP (2) CRNP (3) EB | (1) CRNP (2) EB (3) CRHP | (1) CRNP (2) CRHP (3) EB | (1) EB (2) CRHP (3) CRNP | (1) EB (2) CRNP (3) CRHP
Started | 3 | 4 | 2 | 3 | 2 | 1
Completed | 2 | 1 | 2 | 3 | 2 | 0
Not Completed | 1 | 3 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 1
Period: Washout 1 (14 Days)
Arm/Group | (1) CRHP (2) EB (3) CRNP | (1) CRHP (2) CRNP (3) EB | (1) CRNP (2) EB (3) CRHP | (1) CRNP (2) CRHP (3) EB | (1) EB (2) CRHP (3) CRNP | (1) EB (2) CRNP (3) CRHP
Started | 2 | 1 | 2 | 3 | 2 | 0
Completed | 2 | 1 | 0 | 3 | 1 | 0
Not Completed | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 1 | 0
Period: Intervention 2 (5 Days)
Arm/Group | (1) CRHP (2) EB (3) CRNP | (1) CRHP (2) CRNP (3) EB | (1) CRNP (2) EB (3) CRHP | (1) CRNP (2) CRHP (3) EB | (1) EB (2) CRHP (3) CRNP | (1) EB (2) CRNP (3) CRHP
Started | 2 | 1 | 0 | 3 | 1 | 0
Completed | 2 | 1 | 0 | 3 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 2 (14 Days)
Arm/Group | (1) CRHP (2) EB (3) CRNP | (1) CRHP (2) CRNP (3) EB | (1) CRNP (2) EB (3) CRHP | (1) CRNP (2) CRHP (3) EB | (1) EB (2) CRHP (3) CRNP | (1) EB (2) CRNP (3) CRHP
Started | 2 | 1 | 0 | 3 | 1 | 0
Completed | 2 | 1 | 0 | 3 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 3 (5 Days)
Arm/Group | (1) CRHP (2) EB (3) CRNP | (1) CRHP (2) CRNP (3) EB | (1) CRNP (2) EB (3) CRHP | (1) CRNP (2) CRHP (3) EB | (1) EB (2) CRHP (3) CRNP | (1) EB (2) CRNP (3) CRHP
Started | 2 | 1 | 0 | 3 | 1 | 0
Completed | 2 | 1 | 0 | 3 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (1) CRHP (2) EB (3) CRNP | (1) CRHP (2) CRNP (3) EB | (1) CRNP (2) EB (3) CRHP | (1) CRNP (2) CRHP (3) EB | (1) EB (2) CRHP (3) CRNP | (1) EB (2) CRNP (3) CRHP | Total
Number analyzed (Participants) | 3 | 4 | 2 | 3 | 2 | 1 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 2 | 3 | 2 | 1 | 15
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.3 (3.2) | 19.5 (0.6) | 21 (0) | 25.3 (3.8) | 27 (1.4) | 21 (0) | 22.3 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 4 | 2 | 3 | 2 | 1 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 2 | 3 | 2 | 1 | 15
Percentage Body Fat [Mean (Standard Deviation); unit: % body fat] | 17.9 (5.2) | 13.4 (4.4) | 12 (0.1) | 18 (1.7) | 19.2 (1.8) | 15 (0) | 15.9 (4.0)
Aerobic Fitness (VO2max) [Mean (Standard Deviation); unit: mL/kg/min] | 43.4 (2.1) | 46.7 (5.2) | 47.1 (6.5) | 41.0 (10.4) | 41.6 (5.0) | 42.3 (0) | 43.6 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting Metabolic Rate
Time Frame: Baseline and day 6
Measure: Mean (Standard Error); unit: kcal change
Arm/Group | Caloric Restriction and High Protein | Caloric Restriction and Normal Protein | Energy Balance
Number analyzed (Participants) | 7 | 7 | 7
kcal change | -63.4 (58.2) | -77.6 (100.1) | -47.4 (41.7)

2. Primary Outcome: Change in Circulating IGF-1
Time Frame: Baseline and day 6
Population: All participants completing each condition.
Measure: Mean (Standard Error); unit: mol/L change
Arm/Group | Caloric Restriction and High Protein | Caloric Restriction and Normal Protein | Energy Balance
Number analyzed (Participants) | 7 | 7 | 7
mol/L change | -2.3195714 (1.144509) | -0.2107857 (2.369683) | -1.1142857 (1.628160)

3. Primary Outcome: Change in Marker of Bone Formation (P1NP)
Time Frame: Baseline and day 6
Population: Participants who completed all conditions.
Measure: Mean (Standard Error); unit: % change
Arm/Group | Caloric Restriction and High Protein | Caloric Restriction and Normal Protein | Energy Balance
Number analyzed (Participants) | 7 | 7 | 7
% change | 3.73 (16.82) | 4.80 (19.78) | -3.24 (8.95)

4. Primary Outcome: Change in Marker of Bone Resorption (CTx)
Time Frame: Baseline and day 6
Measure: Mean (Standard Error); unit: % change
Arm/Group | Caloric Restriction and High Protein | Caloric Restriction and Normal Protein | Energy Balance
Number analyzed (Participants) | 7 | 7 | 7
% change | 0.24 (5.56) | 6.93 (16.51) | -8.34 (10.41)

5. Secondary Outcome: Change in Body Weight
Time Frame: Baseline and day 6
Measure: Mean (Standard Error); unit: kg
Arm/Group | Caloric Restriction and High Protein | Caloric Restriction and Normal Protein | Energy Balance
Number analyzed (Participants) | 7 | 7 | 7
kg | -2.3 (0.5) | -2.1 (0.3) | -0.0 (0.3)

6. Secondary Outcome: Change in Body Fat Percentage
Time Frame: Baseline and day 6
Population: Due to equipment errors, n = 5 participants had complete body composition data for all conditions.
Measure: Mean (Standard Error); unit: % change
Arm/Group | Caloric Restriction and High Protein | Caloric Restriction and Normal Protein | Energy Balance
Number analyzed (Participants) | 5 | 5 | 5
% change | -0.94 (0.23) | -0.23 (0.41) | -0.08 (0.53)

7. Secondary Outcome: Change in Aerobic Fitness (VO2peak)
Description: Analyzed in L/min rather than mL/kg/min to remove influence of weight loss.
Time Frame: Baseline and day 6
Population: n = 1 participants had data missing from post-testing in one condition due to equipment failure so their data for the other conditions was removed
Measure: Mean (Standard Error); unit: L/min change
Arm/Group | Caloric Restriction and High Protein | Caloric Restriction and Normal Protein | Energy Balance
Number analyzed (Participants) | 6 | 6 | 6
L/min change | 0.25 (0.08) | 0.01 (0.06) | 0.01 (0.12)

8. Secondary Outcome: Change in Perceived Hunger
Description: Perceived hunger will be assessed using 0-100 visual analog scales. In this case, 100 means maximum hunger while 0 means minimal hunger.
Time Frame: Baseline and day 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Caloric Restriction and High Protein | Caloric Restriction and Normal Protein | Energy Balance
Number analyzed (Participants) | 7 | 7 | 7
units on a scale | 18.4 (5.2) | 27.3 (11.9) | 10.3 (2.9)

ADVERSE EVENTS:
Time Frame: During the course of the entire study (~1.5 years).
Arm/Group | Caloric Restriction and High Protein | Caloric Restriction and Normal Protein | Energy Balance
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/11 | 0/9 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caloric Restriction and High Protein (N=11) | Caloric Restriction and Normal Protein (N=9) | Energy Balance (N=9)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT02945410/Prot_SAP_000.pdf